CLINICAL TRIAL: NCT05305612
Title: Strategy To Optimize PeriproCeduraL AnticOagulation in Structural Transseptal Interventions
Brief Title: Optimal PeriproCeduraL AnticOagulation in Structural Transseptal Interventions
Acronym: STOP CLOT
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Collaborators: Medical Research Agency, Poland (Other Government); Soft Communication, Poland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABM/2020/1/00002
Record Dates: First submitted 2022-03-14; First posted 2022-03-31 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-10

CONDITIONS: Mitral Regurgitation; Atrial Fibrillation; Anticoagulation
MeSH Terms: conditions — Mitral Valve Insufficiency; Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to:
  Early unfractionated heparin administration. The iv. bolus of UFH (100Units/kg) will be given after obtained femoral vein access and at least 5 minutes prior to the start of the TSP.
  Late unfractionated heparin administration. The iv. bolus of UFH (100Units/kg) will be given immediately after TSP, defined as the introduction of transseptal sheath into the left atrium.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be conducted by blinded and unblinded staff. The participants, investigators, care provider and outcome assessors will be blinded. However, in every center the dedicated unblinded study nurse will randomize the patient and prepare two syringes either with saline or UFH. The syringes will be labeled with number 1 and number 2 and will be provided to the anestesiologist taking care of patient during the procedure. The injection from syringe nr 1 will be administered after obtaining the venous access and 5 minutes before the start of TSP. The injection from syringe nr 2 will be administered after TSP defined as introduction of trans-septal sheath into the left atrium. The unblinding nurse responsible for the randomization procedure and preparation of syringe nr 1 and syringe nr 2 and will be not involved in any other procedures or care of the patients enrolled into the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early UFH administration (Experimental): The iv. bolus of UFH (100Units/kg) will be given after obtained femoral vein access and at least 5 minutes prior to the start of the TSP.
  Interventions: Other: early anticoagulation
- Late UFH administration (Active Comparator): The iv. bolus of UFH (100Units/kg) will be given immediately after TSP, defined as the introduction of transseptal sheath into the left atrium.
  Interventions: Other: late anticoagulation

INTERVENTIONS:
Other: early anticoagulation — Anticoagulation prior to transseptal puncture
  Arms: Early UFH administration
Other: late anticoagulation — Anticoagulation after transseptal puncture
  Arms: Late UFH administration

SUMMARY:
The transcatheter edge to edge mitral valve repair (TEER) and left atrial appendage closure (LAAC) are the interventional cardiology procedures that require periprocedural anticoagulation with unfractionated heparin (UFH). The UFH is administered either before or immediately after transseptal puncture, at the discretion of the operator

The aim of the study is to establish the optimal timing of initiation of periprocedural anticoagulation in patients undergoing structural heart interventions requiring transseptal puncture (TEER and LAAC), Patients who undergo TEER implantation or LAAC procedure will be randomized to two groups:

1. Early UFH administration. The iv. bolus of UFH (100Units/kg) will be given after obtained femoral vein access and at least 5 minutes prior to the start of the TSP.
2. Late UFH administration. The iv. bolus of UFH (100Units/kg) will be given immediately after TSP, defined as the introduction of transseptal sheath into the left atrium.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years
2. Planned TEER procedure or left atrial appendage closure
3. The patient is willing to sign informed consent and comply will all study procedure

Exclusion Criteria:

1. Women who are pregnant or breastfeeding and those women of childbearing potential who do not agree to use at least two contraceptive measures (oral contraception, mechanical contraception, approved contraceptive implants, intrauterine device, tubal ligation). The criterion does not apply to women who have been postmenopausal for at least 2 years prior to study enrollment (defined as at least one year without menstrual periods) or underwent surgical sterilization procedure. All eligible women who are younger than 55 years must have negative pregnancy test within 24 hours prior to randomization.
2. Congenital or acquire bleeding disorders (i.e.diagnosed thrombophilia, bleeding diathesis, thrombocyopenia with platelet count <50 thousand/ml, INR elevated >1.5 in the last test prior to randomization)
3. INR > 1.5 within 24 hours prior to the procedure in patients chronically treated with vitamin K antagonists. (applies to the last INR value prior to randomization)
4. Last dose of new oral anticoagulant < 48 hours prior to the procedure (assessed at randomization)
5. Last dose of low molecular weight heparin <12 hours prior to the procedure (assessed at randomization)
6. Contraindications to MR imaging (i.e. claustrophobia, ferromagnetic intraocular foreign boddies, ferromagnetic metalic prostheses)
7. Implanted cardiac devices for electrotherapy if:

   * device has epicardial leads
   * left disconnected leads or non-functional or damaged devices
   * device implanted within abdominal wall
   * the patient is pacemaker dependant (lack of escape rhytm >30/min)
   * the device was implanted or exchanged within 6 weeks prior to the MR examination
   * device mulfunction identified during the control performed prior to the MR examination, that in the opinion of electrophysiologist team may impact the safety of MR imaging
   * low voltage of the device battery - the battery on the examination day should have at least 20% of the voltage value between the nominal value and elective replacement indicator (ERI) value, or the expected battery life calculated by the device should equal or exceed one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2022-03-13 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
1. MACCE 2. Intraprocedural fresh thrombus formation in the right or left atrium as assessed with periprocedural transsesophageal echocardiography 3. Occurrence of new ischemic lesions with diameter ≥4 mm in brain MR performed 2-5 days after procedure | Within 30 days from the index procedure
  Major adverse cardiac and cerebrovascular events (MACCE) will include: death, stroke, TIA, peripheral embolization, myocardial infarction within 30 days from the index procedure.

SECONDARY OUTCOMES:
Moderate and severe bleeding complications (BARC 2-5) including cardiac tamponade requiring intervention during the index hospitalization | during the hospitalization related to the index procedure but up to 30 days from randomization
Intraprocedural fresh thrombus formation in the right of left atrium as assessed with periprocedural transsesophageal echocardiography | during index procedure
Occurrence of new ischemic brain lesion in the MR examination performed within 2-5 days post index procedure. | within 2-5 days post index procedure
Major adverse cardiac and cerebrovascular events (death, stroke, TIA, peripheral embolization, myocardial infarction) within 30 days from the index procedure. | within 30 days from index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jerzy Pręgowski, MD, PhD, Principal Investigator — National Institute of Cardiology
Locations (5):
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne Gdański Uniwersytet Medyczny, Gdansk
  - Górnośląskie Centrum Medyczne im. Leszka Gieca Śląskiego Uniwersytetu Medycznego, Katowice
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie, Lublin
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
to be defined
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD sharing will be considered after study completion and publication of the results.
Access Criteria: to be defined

REFERENCES:
- [Derived] Pregowski J, Pracon R, Mioduszewska A, Skowronski J, Sondergaard L, Mintz GS, Capodanno D, Kim SW, De Baker O, Wacinski P, Wojakowski W, Rdzanek A, Grygier M, Chmielecki M, Franco LN, Stoklosa P, Firek B, Marczak M, Milosz B, Chmielak Z, Demkow M, Witkowski A. Strategy to optimize PeriproCeduraL AnticOagulation in structural transseptal interventions: Design and rationale of the STOP CLOT trial. Am Heart J. 2024 May;271:68-75. doi: 10.1016/j.ahj.2024.02.015. Epub 2024 Feb 22. PMID 38401649